CLINICAL TRIAL: NCT05788497
Title: Multicentre, Double-blind, Randomised Clinical Trial to Evaluate and Compare the Efficacy and Safety of Hemorrane Plus (Hemorrane® + Benzocaine) With Hemorrane® and With Placebo in Patients With Uncomplicated Haemorrhoids
Brief Title: Efficacy and Safety of Hemorrane Plus Versus Hemorrane and Versus Placebo in Patients With Uncomplicated Haemorrhoids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Recruitment failure
Sponsor: Faes Farma, S.A. (Industry)
Collaborators: Dynamic Science S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEMP-0119/ES
Record Dates: First submitted 2023-03-15; First posted 2023-03-29 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Haemorrhoids Without Complication
Keywords: Haemorrhoids; Haemorrhoids without complication
MeSH Terms: conditions — Hemorrhoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hemorrane® Plus (Experimental): Daily application of Hemorrane Plus (Hemorrane® + benzocaine) 10 mg/g rectal ointment + 30 mg/g benzocaine for 7 days.
  Interventions: Drug: Hemorrane plus
- Hemorrane® (Active Comparator): Daily application of Hemorrane 10 mg/g rectal ointment for 7 days.
  Interventions: Drug: Hemorrane
- Placebo (Placebo Comparator): Daily application of placebo for 7 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Hemorrane plus — Hemorrane 10 mg/g rectal ointment + 30 mg/g benzocaine
  Arms: Hemorrane® Plus
Drug: Hemorrane — Hemorrane 10 mg/g rectal ointment
  Arms: Hemorrane®
Drug: Placebo — Rectal ointment
  Arms: Placebo

SUMMARY:
This is a Multicentre, double-blind, randomised clinical trial to evaluate and compare the efficacy and safety of Hemorrane Plus (Hemorrane® + benzocaine) with Hemorrane® and with placebo in patients with uncomplicated haemorrhoids.

ELIGIBILITY:
Inclusion Criteria:

1. Over 18s and both sexes.
2. Voluntary signing of informed consent.
3. Diagnosis of uncomplicated haemorrhoids: grade I or II non-thrombosed external, mixed, or internal haemorrhoids.
4. VAS of pain ≥ 5 points.
5. VAS of pruritus and stinging/burning ≥ 5 points (for each one).
6. Commitment to comply with the hygienic-dietary measures established for the general management of haemorrhoids.
7. Negative urine pregnancy test (women of childbearing age, if applicable).
8. Patients with adequate understanding of the study and ability to perform the procedures independently.

Exclusion Criteria:

1. History of hypersensitivity to any of the active ingredients or components of the investigational products, as well as hypersensitivity to other local anaesthetics derived from para-aminobenzoic acid (PABA), parabens, or paraphenylenediamine (for example, hair dyes, henna tattoos).
2. Use of topical haemorrhoid medications or other topical agents for the anorectal area less than 48 hours before the start of the study (Visit 1, day 1).
3. Haemorrhoidal surgery that is scheduled between Visit 1 (day 1) and the follow-up visit Visit 3 (day 15±2).
4. Diagnosis of grade III or IV thrombosed external or internal haemorrhoids.
5. Medical history of anaemia, and/or current diagnosis of cardiac or pulmonary disease, shock, sepsis, acidosis, or genetic predisposition (NADH-cytochrome b5 reductase deficiency, glucose-6-phosphate dehydrogenase deficiency, and haemoglobin M disease); that include risk factors for methemoglobinemia.
6. Documented diagnosis of active tuberculosis.
7. Active bleeding haemorrhoids.
8. Presence of pain, stinging/burning, pruritus, anorectal bleeding or rectal bleeding for causes other than haemorrhoidal disease.
9. Presence of bacterial, viral, and/or fungal infections in the perianal area.
10. History of pancreatic pathology that may require performance of a bentiromide diagnostic test.
11. Use of any of the prohibited concomitant medications (sulfonamides, cholinesterase inhibitors, ester or prilocaine-type local anaesthetics, sodium nitrite, neurotoxic insecticides (topical malathion), aminosalicylic acid, suxamethonium, antiarrhythmics, monoamine oxidase inhibitors, tricyclic antidepressants, and PABA derivatives) less than one week prior to the start of the study (Visit 1, Day 1), or throughout the study.
12. Use of any hair dye, including those containing paraphenylene-diamine during the study, from Visit 1 (Day 1) to the follow-up Visit 3 (Day 15 ± 2).
13. Any other circumstance considered by the investigator to prevent adequate follow-up and/or adequate evolution of the response to the study treatments.
14. Pregnant women, those planning an upcoming pregnancy or breast-feeding.
15. Women of childbearing age who do not agree to take the pregnancy test and use valid contraceptive methods during the study and until the end of the use of the investigational treatment. The following are considered valid contraceptive methods: combined hormonal oral, intravaginal or transdermal contraceptives (oestrogen and progesterone), oral, injectable or implantable progesterone-based hormonal contraceptives, intrauterine device (IUD), hormone-releasing intrauterine device, bilateral tubal occlusion, vasectomised partner (as long as they are the only sexual partner of the participating patient and that the success of the intervention has been medically confirmed), or sexual abstinence (abstaining from heterosexual intercourse during the treatment period). The investigator is responsible for determining whether the patient has an appropriate contraceptive method for her participation in the study.
16. Fertile men who use condoms or have had a vasectomy (as long as the success of the intervention has been medically confirmed), or who practise abstinence (abstinence from heterosexual sexual relationships during the treatment period). The investigator is responsible for determining whether the patient has an appropriate contraceptive method for their participation in the study.
17. Patients who have had active cancer in the last five years.
18. Patients who have received an investigational drug (including vaccines) or who have used an invasive medical device in the last 30 days prior to the start of the screening phase or who are currently participating in another clinical trial.
19. Patients who have a family or professional relationship with the research team participating in the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2024-01-04 (Actual); Study Completion 2024-01-04 (Actual)

PRIMARY OUTCOMES:
Percentage of responders at T156h +30 min (day 7 hour 12 + 30min) compared to T0 (day 1 hour 0), for Hemorrane Plus and placebo; as well as the percentage of responders within 30 minutes after the application of Hemorrane Plus and Hemorrane®. | 7 days 12 hours 30 min
  Responders are defined as those patients with a decrease of two or more points out of ten on the Visual Analogue Scale (VAS) of pain (assessed by the patient).

SECONDARY OUTCOMES:
Percentage of responders at T156h +30 min (day 7 hour 12 + 30 min) compared to T0 (day 1 hour 0), for Hemorrane® Plus versus placebo | 7 days 12 hours 30 min
  Responders are defined as those patients with a decrease of two or more points out of ten on the Visual Analogue Scale (VAS) of pain (assessed by the patient).
Percentage of responders at T156h +30 min (day 7 hour 12 + 30min) compared to T0 (day 1 hour 0), for Hemorrane Plus and Hemorrane® | 7 days 12 hours 30 min
  Responders are defined as those patients with a decrease of two or more points out of ten on the Visual Analogue Scale (VAS) of pain (assessed by the patient).
Change in the VAS of pruritus (assessed by the patient), at the established times, compared to the baseline value (T0), for the three treatments. | 7 days 12 hours 30 min
  Change in the VAS of pruritus at the established times after the application of te ointment for each of the treatments assessed by the patient using the electronic diary.
Change in the VAS of stinging/burning (assessed by the patient), at the established times, compared to the baseline value (T0), for the three treatments. | 7 days 12 hours 30 min
  Change in the VAS of pruritus at the established times after the application of te ointment for each of the treatments assessed by the patient using the electronic diary.
Evaluation of the mean values of the bleeding episodes recorded (assessed by the investigator) at Visit 1 (Screening and baseline), and at Visit 2 (day 8+1), for the three treatments. | 7 days 12 hours 30 min
  The investigator will ask about bleeding episodes before first application and after finishing the treatment (day 8+1)
Change in the VAS of inflammation (assessed by the investigator) at Visit 2 (day 8+1), compared to baseline (T0), for the three treatments. | 7 days 12 hours 30 min
  The investigator will evaluate the inflammation prior to the application of the ointment and after finishing the treatment (day 8+1)
Change in the patient's quality of life measured with the EQ-5D-5L questionnaire, at Visit 2 (day 8+1) compared to the baseline value at Visit 1 (day 1, T0), for the three treatments | 7 days 12 hours 30 min
  A quality of life questionary will be given to patients for the three treatments before and after the application of the ointment.
Incidence of adverse events (AE) | 7 days 12 hours 30 min
  Incidence of adverse events (AE) for the three treatments
Incidence of topical allergic reactions | 7 days 12 hours 30 min
  Incidence of topical allergic reactions for the three treatments
Description of local tolerability and satisfaction | 7 days 12 hours 30 min
  Description of local tolerability and satisfaction for the three treatments
Percentage of clinically significant changes in haematology, biochemistry, and methaemoglobin analysis compared to baseline. | 15 +/- 2 days
  A blood sample will be obtained before and two weeks after the start of the treatment.
Percentage of patients withdrawn from the study for safety reasons | 7 days 12 hours 30 min

CONTACTS AND LOCATIONS:
Locations (13):
- Spain (13):
  - CAP Can Bou, Castelldefels, Barcelona
  - CAP Corbera de Llobregat, Corbera de Llobregat, Barcelona
  - CAPSBE Les Corts, L'Hospitalet de Llobregat, Barcelona
  - CS Dr. Mendiguchia Carriche, Leganés, Madrid
  - CS Las Fronteras, Torrejón de Ardoz, Madrid
  - CS A Estrada, A Estrada, Pontevedra
  - CS Trinitat, Valencia, Valencia
  - CS Trafalgar, Valencia, Valencia
  - CS Ávila Estación, Ávila
  - CS Montesa, Madrid
  - CS Goya, Madrid
  - CS Fuencarral, Madrid
  - CS General Fanjul, Madrid